CLINICAL TRIAL: NCT07397650
Title: Efficacy and Safety With Early Treatment of Finerenone in Hospitalized Patients With Heart Failure
Acronym: FACILITATE-HF
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Juntendo University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: jRCTs031250369
Record Dates: First submitted 2026-02-02; First posted 2026-02-09 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Acute Heart Failure
MeSH Terms: interventions — finerenone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Finerenone (Experimental): Patients will be randomized 1:1 to either finerenone or placebo.
  Interventions: Drug: Finerenone Oral Tablet
- Placebo (Placebo Comparator): Placebo tablets matching finerenone are administered orally
  Interventions: Drug: Finerenone Placebo

INTERVENTIONS:
Drug: Finerenone Oral Tablet — For participants with an eGFR ≤60 mL/min/1.73 m^2: Starting dose is 10 mg OD and maximum dose 20 mg OD.
  For participants with an eGFR >60 mL/min/1.73 m^2: Starting dose is 20 mg OD and maximum dose 40 mg OD.
  Arms: Finerenone
Drug: Finerenone Placebo — Placebo tablets matching finerenone are administered orally
  Arms: Placebo

SUMMARY:
FACILITATE-HF is a multicenter, randomized, double-blind, placebo-controlled trial designed to determine whether initiation of finerenone during the early phase of hospitalization has beneficial effects in patients with AHF who have left ventricular ejection fraction 40% or more.

ELIGIBILITY:
Patients eligible for inclusion in this study meet all of the following criteria: <br>Inclusion Criteria:

1. Patients ≥18 years of age, male or female<br>
2. Current hospitalization with AHF requiring intravenous loop diuretics or vasodilators during the index admission<br>
3. Patients have to have at least one of new or worsening symptoms due to HF and one of new or worsening physical examination findings due to HF <br> (i) symptom<br> dyspnoea, decreased exercise tolerance, or fatigue<br> (ii) physical examination<br> peripheral edema, increasing abdominal distention or ascites, pulmonary rales/crackles/crepitations, increased jugular venous pressure and/or hepatojugular reflux, S3 gallop, clinically significant or rapid weight gain<br>
4. Patients who are not hemodynamically unstable as defined by meeting the following criteria<br>

   1. Systolic blood pressure ≥100 mmHg and no symptoms of hypotension within 6 hours prior to randomization<br>
   2. No increase in intravenous diuretic dose or intravenous vasodilators within 6 hours prior to randomization with worsening HF symptom<br>
   3. Without cardiogenic shock, no use of inotropes or vasopressors, no use of mechanical circulatory support, not requiring intubation after admission, and not expected to require inotropes, vasopressors, mechanical circulatory support or intubation during the index hospitalization<br>
5. NTproBNP ≥1500 pg/mL or BNP ≥375 pg/mL (For patients treated with ARNI in the previous 4 weeks prior to randomization, only NT-proBNP values should be used)<br>
6. Most recent LVEF ≥40% within the past 1 year <br>
7. Randomization within 24 hours after admission, and drug administration within 36 hours after admission <br>
8. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol<br>
9. Signed informed consent must be obtained prior to participation in the study<br>

Exclusion Criteria:

1. Estimated glomerular filtration rate (eGFR) <25 mL/min/1.73m2 by CKD-EPI Creatinine Equation (2021) at screening<br>
2. Serum/plasma potassium >5.0 mmol/L at screening<br>
3. Patients who cannot receive oral treatment<br>
4. Use of eplerenone, spironolactone, esaxerenone or potassium-sparing diuretic within 30 days before randomization <br>
5. Known hypersensitivity to the study intervention (active substance or excipients)<br>
6. Systemic therapy with potent cytochrome P450 isoenzyme 3A4 (CYP3A4) inhibitors or inducers within 7 days before randomization or is expected to be used during the study period (e.g. itraconazole, ritonavir, indinavir, cobicistat, clarithromycin).<br>
7. Participants who require treatment with more than one ACEI, ARB or angiotensin-receptor neprilysin inhibitor (ARNI) simultaneously<br>
8. Acute heart failure in which other diseases are the main cause of symptoms and signs (chronic obstructive pulmonary disease, anemia, etc.)<br>
9. Patients who are on dialysis including peritoneal dialysis or in whom the initiation of dialysis during the study period<br>
10. Pregnant or lactating female<br>
11. Acute coronary syndrome, pulmonary thromboembolism, stroke, or transient ischemic attack within 90 days before randomization.<br>
12. Have undergone the following therapeutic intervention within 30 days before randomization: cardiovascular surgery (e.g., coronary artery bypass grafting, surgery for valvular heart disease, transcatheter aortic valve implantation, percutaneous coronary intervention, percutaneous edge-to-edge mitral valve repair, and other types of surgery at the investigator's discretion) and implantation of an implantable defibrillator, or a cardiac resynchronization therapy defibrillator.<br>
13. Heart transplant recipients or patients listed for heart transplantation who are expected to undergo transplantation during the study, patients implanted with an implantable ventricular-assist device, patients expected to require an implantable ventricular-assist device during the study, and patients expected to switch to palliative care during the study.<br>
14. Coronary or valvular heart disease likely to require surgical or percutaneous intervention within the study period (there is no reason to exclude secondary mitral or tricuspid regurgitation due to reduced cardiac function, except for the absence of a plan to perform cardiac surgery or therapeutic catheterization)<br>
15. Secondary cardiomyopathy such as amyloidosis, cardiac sarcoidosis, hemochromatosis, Fabry's disease, chemotherapy induced cardiomyopathy, and muscular dystrophy. Heart failure due to takotsubo cardiomyopathy, obstructive hypertrophic cardiomyopathy, complex congenital heart disease (as determined by the investigator), pericardial constriction, right heart failure in absence of left-sided structural disease<br>
16. Acute cardiac structural abnormalities (e.g., acute mitral regurgitation due to ruptured chordae tendineae and infective endocarditis)<br>
17. Peripartum cardiomyopathy diagnosed within 6 months before randomization.<br>
18. Active myocarditis at randomization.<br>
19. Patients with symptomatic bradycardia or complete atrioventricular block who are being treated with temporary pacemaker implantation at the time of admission, or who are expected to require temporary or permanent pacemaker implantation in the future. Patients who have already been treated with permanent pacemaker implantation do not meet the exclusion criteria<br>
20. Presence of uncontrolled thyroid disease<br>
21. Addison's disease<br>
22. Hepatic insufficiency classified as Child-Pugh C <br>
23. Patients with excessive alcohol intake (15+ drinks/week for men, 8+ drinks/week for women)<br>
24. Any other condition or therapy, which would make the participant unsuitable for this study and will not allow participation for the full planned study period (e.g. active malignancy or other condition limiting life expectancy to less than 12 months)<br>
25. Patients with dementia. If a sub-investigator determines that confirmation of cognitive impairment is necessary, it must be verified that the Mini-Cog score is not less than 4.<br>
26. Participation in another interventional clinical study (e.g. phase 1 to 3 clinical studies) or treatment with another investigational medicinal product within 30 days prior to randomization.Other conditions likely to interfere with the patient's safety or compliance with the protocol<br>
27. Patients deemed unsuitable by the principal investigator or sub investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 550 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
A hierarchical composite endpoint of death and worsening heart failure | Up to 12 weeks
  A hierarchical composite endpoint consisting of death, worsening HF during hospitalization, HF rehospitalization, worsening HF after discharge requiring IV diuretic or sustained intensification of oral therapy, and change in N-terminal pro-B-type natriuretic peptide levels at 12 weeks as assessed using a win ratio

SECONDARY OUTCOMES:
All-cause death | Up to 12 weeks
Cardiovascular death | Up to 12 weeks
Worsening HF during hospitalization | During hospitalization
HF rehospitalization | Up to 12 weeks
Worsening HF after discharge requiring IV diuretic or sustained intensification of oral therapy | Up to 12 weeks
NT-proBNP change from baseline to 12 weeks | Up to 12 weeks
Kansas City Cardiomyopathy Questionnaire - Total Symptom Score from baseline to 12 weeks | Up to 12 weeks
  Kansas City Cardiomyopathy Questionnaire - Total Symptom Score from baseline to 12 weeks. The scores range from 0 to 100, with higher scores indicating fewer symptoms and physical limitations.
Urine output from randomization to 48 hours | Up to 48 hours
Change in patient dyspnea in the supine position assessed by a visual analogue scale from randomization to discharge and to 12 weeks | Up to 12 weeks
  Change in patient dyspnea in the supine position assessed by a visual analogue scale from randomization to discharge and to 12 weeks. The scores range from 0 to 100, with 100 being the best possible score.
Symptomatic atrial fibrillation up to discharge and up to 12 weeks | Up to 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yuya Matsue, MD, Principal Investigator — Department of Cardiovascular Biology and Medicine, Juntendo University Graduate School of Medicine
Locations (21):
- Japan (21):
  - Chita Peninsula General Medical Center, Handa, Aichi-ken
  - Japanese Red Cross Aichi Medical Center Nagoya Daini Hospital, Nagoya, Aichi-ken
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - National Center for Geriatrics and Gerontology, Ōbu, Aichi-ken
  - Toyota Kosei Hospital, Toyota, Aichi-ken
  - Ehime University Hospital, Tōon, Ehime
  - Japanese Red Cross Fukuoka Hospital, Fukuoka, Fukuoka
  - Iizuka Hospital, Iizuka, Fukuoka
  - Gunma Prefectural Cardiovascular Center, Maebashi, Gunma
  - Gunma University Hospital, Maebashi, Gunma
  - NHO Takasaki General Medical Center, Takasaki, Gunma
  - Hokkaido Cardiovascular Hospital, Sapporo, Hokkaido
  - Kitasato University Hospital, Sagamihara, Kanagawa
  - Kindai University Hospital, Sakai, Osaka
  - National Cerebral and Cardiovascular Center, Suita, Osaka
  - The University of Osaka Hospital, Suita, Osaka
  - Saitama Medical Center, Kawagoe, Saitama
  - Juntendo University Shizuoka Hospital, Izunokuni, Shizuoka
  - Chutoen General Medical Center, Kakegawa, Shizuoka
  - Osaka General Medical Center, Osaka
  - Juntendo University Hospital, Tokyo

IPD SHARING:
Plan to Share IPD: Undecided